CLINICAL TRIAL: NCT05153304
Title: A Phase I/II Study of Personalized Immunotherapy in Adults With Upper Gastrointestinal Tract Cancers
Brief Title: Personalized Immunotherapy in Adults With Upper Gastrointestinal Tract Cancers
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: funding
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Ezra Cohen, Physician, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCV-001
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Cancer of Gastrointestinal Tract
Keywords: cancer; gastrointestinal; immunotherapy; personalized cancer vaccine; nivolumab; neoantigen; vaccine
MeSH Terms: conditions — Gastrointestinal Neoplasms; Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- anti-PD1 and personalized vaccine (Experimental)
  Interventions: Biological: personalized vaccine; Drug: Nivolumab

INTERVENTIONS:
Biological: personalized vaccine — Vaccine will be constructed for each subject that express multiple candidate tumor-derived neoantigens.
Drug: Nivolumab — 3mg/kg nivolumab will be administered intravenous (IV) infusion every 3 weeks for 4 doses. After 4 doses, 480 mg nivolumab will be administered intravenous (IV) infusion every 4 weeks.
  Other Names: Opdivo

SUMMARY:
The purpose of this study is to determine if it is possible to make and safely administer a 'personalized' cancer vaccine for people diagnosed with an upper gastrointestinal tract cancer.

DETAILED DESCRIPTION:
The purpose of this study is to determine if it is possible to make and safely administer a 'personalized' cancer vaccine for people diagnosed with an upper gastrointestinal tract cancer.

It is known that cancer has mutations (changes in genetic material) that are specific to an individual person and their tumor. These mutations can cause the tumor cells to produce proteins that are different from the body's normal, healthy cells. The study will use a sample of your tumor to create a vaccine against it, with the idea being that the study vaccine will "teach" the body's immune system to recognize and attack the cancer cells. The study will examine the safety of the study vaccine when given at several time points and will examine your blood for signs that the study vaccine causes the immune system to respond.

The personalized cancer vaccine will be given alone or in combination with nivolumab. Nivolumab is a drug that blocks certain proteins on cells that help to keep immune responses in check. In a healthy person, this keeps the immune system from attacking healthy cells and tissues, but cancer cells use these proteins to keep the immune system from killing cancer cells and tumors. When these proteins are blocked, the check on the immune system is removed and immune cells may be able to recognize and kill cancer cells.

This personalized cancer vaccine is considered experimental because it is not approved by the US Food & Drug Administration (FDA) as a treatment for cancer.

The combination of nivolumab and the personalized cancer vaccine is experimental and is not FDA approved.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented gastroespohageal or gastric adenocarcinoma.
* Measurable disease as defined by RECIST 1.1
* Adequate organ function
* Women of child-bearing potential and men with partners of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence)

Exclusion Criteria:

* Currently receiving or has received another anti-cancer therapy within 4 weeks prior to first dose of vaccine study treatment.
* Currently receiving or has received PD1/PDL1 inhibitor immunotherapy within 4 weeks prior to first dose of study treatment.
* Received an investigational agent within 28 days prior to the first dose of study drug.
* Untreated brain metastases; individuals with treated and stable metastases are eligible. Eligible subjects should have recovered from the acute effects of radiation therapy or surgery prior to study entry, have discontinued corticosteroid treatment for brain metastases for at least 4 weeks and are neurologically stable for 8 weeks (confirmed by MRI) prior to administration of experimental therapy
* Has known history of Human Immunodeficiency Virus (HIV).
* Received a diagnosis of hepatitis B or hepatitis C for which there is no clear evidence of natural immunity, immunity subsequent to vaccination, or successful eradication of the virus following antiviral therapy (individuals who are hepatitis C antibody positive may be enrolled if negative viral load confirmed).
* History of autoimmune disease including: inflammatory bowel disease (including ulcerative colitis and Crohn's Disease), rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus, autoimmune vasculitis (e.g. Wegener's granulomatosis); central nervous system or motor neuropathy considered of autoimmune origin (e.g. Guillain-Barré syndrome, myasthenia gravis, multiple sclerosis). Individuals with vitiligo, Sjogren's Syndrome, interstitial cystitis, Graves' or Hashimoto's Disease, celiac disease, DM1, or hypothyroidism stable on hormone replacement will be allowed with Study Medical Monitor's approval.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* History of receiving a solid organ transplant or allogeneic bone marrow transplant.
* Major surgical procedure within 28 days prior to the first dose of study drug.
* If female, pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Quantitative frequency of TCR | 1 year
Treatment-related Adverse Events | 1 year

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 1 year
Overall Survival | 1 year
Overall Response | 1 year
Duration of response | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ezra Cohen, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States